CLINICAL TRIAL: NCT01428154
Title: An Open-label, Single-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Darbepoetin Alfa in Paediatric Subjects From Birth to Less Than 1 Year of Age With Anemia Due to Chronic Kidney Disease
Brief Title: Study to Evaluate Darbepoetin Alfa in Pediatric Subjects With Anemia Due to Chronic Kidney Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty in recruitment. PDCO in the Day 30 summary report agrred to remove the PK study in children <1 year of age.
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20090302
Record Dates: First submitted 2011-09-01; First posted 2011-09-02 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Anemia; Chronic Kidney Disease
Keywords: paediatric; dialysis; CKD; pediatric
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Darbepoetin alfa (Experimental)
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa — A single 1.5 μg/kg subcutaneous (SC) dose administration on day 1
  Other Names: Aranesp

SUMMARY:
The purpose of this study is to find out more about darbepoetin alfa in children less than 1 year of age with anemia (a decrease in red blood cells) due to kidney failure. This study will see if darbepoetin alfa is safe and well tolerated and whether it causes any side effects by taking blood samples and checking vital signs (heart rate, body temperature, and blood pressure tests) at specific times throughout the study. In addition, the study will evaluate the amount of darbepoetin alfa in the blood over time and look at special markers in the blood to evaluate how darbepoetin alfa works on anemia.

Darbepoetin alfa is approved by the United States Food and Drug Administration (FDA) and European Medicines Agency (EMA) for use in adults, but not for all ages of pediatric subjects. Therefore, studies need to be conducted in pediatric subjects (children) to determine the appropriate dose to use in younger children.

ELIGIBILITY:
Inclusion Criteria:

* Girls and boys between birth and < 1 year of age at the time of enrollment
* Body weight ≥ 3 kg at screening and enrollment
* Diagnosis of chronic kidney disease stage 3 to 5 with an estimated Glomerular Filtration Rate < 60 mL/min/1.73m2 without dialysis using the updated Schwartz Equation at screening; OR on dialysis at screening
* Hemoglobin ≤ 9.0 g/dL within 7 days prior to enrollment
* Transferrin saturation ≥ 20% at screening

Exclusion Criteria:

* Premature girls and boys (< 37 weeks of gestation, counting from the first day of the mother's last menstrual period)
* Peritoneal dialysis subjects with an episode of peritonitis within 30 days prior to enrollment
* History of cardiovascular events or thromboembolism
* History of upper or lower gastrointestinal bleeding
* History of seizures
* Active liver disease or history of liver disease
* Uncontrolled hypertension defined as stage 2 hypertension or greater. This is defined as a systolic or diastolic blood pressure value greater than the 99th percentile + 5 mmHg for a subject's age
* Major surgery 12 weeks prior to enrollment
* Red blood cell transfusions 12 weeks prior to enrollment
* Use of any erythropoiesis-stimulating agent within 12 weeks prior to enrollment
* Currently receiving antibiotic therapy for systemic infection within 4 weeks prior to enrollment
* Current or prior use of immunosuppressants (excluding low-dose corticosteroids, defined as ≤ 0.5 mg/kg per day prednisone or equivalent for ≤ 5 days)
* Subject is receiving a dose higher than 0.5 mg/kg per day of prednisone (or equivalent dose of another corticosteroid) for > 5 days within 4 weeks prior to enrollment
* Receiving or has received any investigational drug (or is currently using an investigational device) within the 30 days or 5 half-lives (whichever is longer) prior to enrollment
* Subject has known hypersensitivity to darbepoetin alfa, r-HuEPO, or to any of the excipients

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with clinically significant changes in physical examinations, laboratory safety tests, and vital signs | Assessed over 29 days
Number of subjects with treatment-emergent adverse events | Assessed over 29 days

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) of darbepoetin alfa | Assessed predose and at 6, 24, 48, 72, and 168 hours postdose
Time at which maximum concentration is observed (Tmax) of darbepoetin alfa | Assessed predose and at 6, 24, 48, 72, and 168 hours postdose
Area under the concentration curve (AUC) of darbepoetin alfa | Assessed predose and at 6, 24, 48, 72, and 168 hours postdose
Terminal half-life (t½) of darbepoetin alfa | Assessed predose and at 6, 24, 48, 72, and 168 hours postdose
Clearance (CL) of darbepoetin alfa | Assessed predose and at 6, 24, 48, 72, and 168 hours postdose
Change in reticulocytes | Assessed from baseline to day 8
Change in reticulocytes | Assessed from baseline to day 29
Change in hemoglobin concentration | Assessed from baseline to day 8
Change in hemoglobin concentration | Assessed from baseline to day 29
Change in iron | Assessed from baseline to day 29
Change in ferritin | Assessed from baseline to day 29
Change in transferrin saturation | Assessed from baseline to day 29

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com